CLINICAL TRIAL: NCT02064634
Title: A Multicenter, Comparative, Open Label, Prospective Observational Study on Discontinuation of Medication Due to Gastrointestinal Adverse Effects for the Patients Being Treated for Osteoarthritis With Anti-inflammatory Analgesic Drug
Brief Title: A Prospective Observational Study on Discontinuation of Medication of Shinbaro Capsule
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Other Study IDs: GCSB_OS
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Shinbaro Capsule; Celecoxib; Osteoarthritis; GCSB-5; Discontinuation rate; Gastrointestinal adverse event; NSAIDs; OASIS
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Shinbaro (only)
- Celecoxib (only)
- Shinbaro + NSAIDs
- Shinbaro + Celecoxib

SUMMARY:
This study investigates how gastrointestinal toxicity affects discontinuation of medication given to patients with osteoarthritis in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 20- year-old patients diagnosed with osteoarthritis
* Within 2 weeks prior to participation, not taken anti-inflammatory analgesic drug such as the Shinbaro Capsule, Celecoxib Capsule and NSAIDs(non-steroidal anti-inflammatory drugs)
* Written consent form voluntarity

Exclusion Criteria:

* Diagnosed with disease that may affect measurement of efficacy clinically
* Diagnosed with clinically significant phycological disorder, and taking medication
* Participated in a clinical trial within 4 weeks
* Pregnant or lactating woman
* History of malignant disease within the previous 5 years
* Patients who seem not to participate in the study at investigator's discretion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis being treated with anti-inflammatory analgesic drug at general hospitals and clinics in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 6700 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate due to gastrointestinal adverse effects | up to 12 weeks

SECONDARY OUTCOMES:
Rate of medication discontinuation recorded as lack of efficacy | up to 12 weeks
  Number of participants discontinued from medication due to lack of efficacy
Rate of medication discontinuation | up to 12 weeks
  Number of participants discontinued from medication
Discontinuation rate due to adverse events | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Sonpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided